CLINICAL TRIAL: NCT06518772
Title: The Effect of Hot Perfoming on the Soles of the Feet in the First Stage of Labor on Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, HATİCE YEŞİLKAYA, Nurse, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: cumhuriyetuniv
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy Related
Keywords: Labor pain, Birth satisfaction, Midwifery, Heat Application
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The application procedure started with the application of hot gel packets at a temperature of 40-42°C to the soles of the feet of the women in the intervention group for 20 minutes when cervical dilation reaches 5 cm.The first Visual Analog Scale (VAS) evaluation was conducted after the application. Conduction is followed by more evaluations at the 25th (5 minutes after the application), 35th (15 minutes after the application), and 50th minute (30 minutes after the application). These applications were repeated every hour until cervical dilation reached 10 cm. The applicatilon procedure has been stopped after cervical dilation reached 10 cm.
  Interventions: Other: hot application
- Control (No Intervention): The control group received routine service and VAS at the same times.

INTERVENTIONS:
Other: hot application — The application procedure started with the application of hot gel packets at a temperature of 40-42°C to the soles of the feet of the women in the intervention group for 20 minutes when cervical dilation reaches 5 cm.
  Arms: Intervention

SUMMARY:
This research was conducted to determine the effect of applying heat to the soles of the feet during the active phase (5-10 cm dilation) of the first stage of labor. It is a randomized controlled experimental study. In the intervention group, hot gel packs with a temperature of 40-42°C were applied to the soles of the feet for 20 minutes when the cervical dilation was 5 cm. These applications were repeated in the same manner at one-hour intervals until the cervical dilation reached 10 cm. The procedure was terminated when the cervical dilation reached 10 cm. Routine services were applied to the control group. Data were collected using a personal information form, Partograph form, APGAR score, Visual Analog Scale (VAS), and Birth Satisfaction Scale Short Form (BSS-SF)

DETAILED DESCRIPTION:
This research was conducted to determine the effect of applying heat to the soles of the feet during the active and transition phase (4-10 cm dilation) of the first stage of labor. The research is a randomized controlled experimental study and is conducted in Sivas Cumhuriyet University Practice and Research Hospital Maternity Unit. When the sample size was taken as α = 0.05 and β = 0.10 and 1-β = 0.90 to represent the population in the research, there were 30 individuals in each group and the power of the test was found to be P = 0.90640. The application procedure started with the application of hot gel packets at a temperature of 40-42°C to the soles of the feet of the women in the intervention group for 20 minutes when cervical dilation reaches 5 cm. The first Visual Analog Scale (VAS) evaluation was conducted after the application. Conduction is followed by more evaluations at the 25th (5 minutes after the application), 35th (15 minutes after the application), and 50th minute (30 minutes after the application). These applications were repeated every hour until cervical dilation reached 10 cm. The applicatilon procedure has been stopped after cervical dilation reached 10 cm. The control group received routine service and VAS at the same times. Data were collected with personal information form, Partograph form, APGAR score, Visual Analog Scale (VAS) and Birth Satisfaction Scale Short Form (BSS-R) Wilcoxon test, Mann Whitney U test, Chi-square test, Exact test, Friedman test, t test were used to evaluate the data. The data error level was accepted as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 1. The pregnant woman must be 19 years or older 2. 38-42. being in the gestational age, 3. Having a singleton pregnancy, 4. The fetus is in a vertex position, 5. Cervical dilatation is 5 cm. to be, 6. Not having a diagnosed chronic physical disease, 7. Not having a diagnosed psychiatric disease, 8. Absence of risky pregnancy and birth, 9. There is no abnormality in the fetus, 10. Being able to speak Turkish and be literate 11. Having a primigravida

Exclusion Criteria:

* Not meeting inclusion criteria

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Because the study was on pregnant women
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Before application
  VAS provides rapid measurement of pain intensity in clinical and laboratory conditions. In VAS, the patient is asked to make a mark on a 10 cm horizontal line showing the current situation. In this study, for pain; Markings are made on a 10 cm horizontal line, one end of which indicates the patient's pain is very good (0 = no pain) and the other end is very bad (10 = most severe).
Visual Analog Scale | 25 minutes after initial pain assessment
  VAS provides rapid measurement of pain intensity in clinical and laboratory conditions. In VAS, the patient is asked to make a mark on a 10 cm horizontal line showing the current situation. In this study, for pain; Markings are made on a 10 cm horizontal line, one end of which indicates the patient's pain is very good (0 = no pain) and the other end is very bad (10 = most severe).
Visual Analog Scale | 35 minutes after initial pain assessment
  VAS provides rapid measurement of pain intensity in clinical and laboratory conditions. In VAS, the patient is asked to make a mark on a 10 cm horizontal line showing the current situation. In this study, for pain; Markings are made on a 10 cm horizontal line, one end of which indicates the patient's pain is very good (0 = no pain) and the other end is very bad (10 = most severe).
Visual Analog Scale | 50 minutes after initial pain assessment
  VAS provides rapid measurement of pain intensity in clinical and laboratory conditions. In VAS, the patient is asked to make a mark on a 10 cm horizontal line showing the current situation. In this study, for pain; Markings are made on a 10 cm horizontal line, one end of which indicates the patient's pain is very good (0 = no pain) and the other end is very bad (10 = most severe).
Birth Satisfaction Scale Short Form | Application of the birth satisfaction scale 2-4 hours after birth
  The scale consists of 10 items and is a Likert type scale. It is scored as "I strongly agree (4 points)", "I agree (3 points)", "I am undecided (2 points)", "I disagree (1 point)", "I strongly disagree (0 points)". 2, 4, 7 of the scale. Items , and 8 are calculated in reverse and the lowest score from the scale is "0" and the highest score is "40". As the score increases, the level of birth satisfaction increases. Scale cut-off scores <13 are low satisfaction, 14-27 are medium satisfaction, >28 are high. The scale has three sub-dimensions: quality of care (3,5,6,10), personal characteristics (8.4) and stress experience (1,2,7,9). The total score that can be obtained from the quality of care sub-dimension is 16. The total score that can be obtained from the personal characteristics sub-dimension is 8 and the total score that can be obtained from the stress experience sub-dimension is 16.

SECONDARY OUTCOMES:
Durations of birth stages with partograph form | during labor
  The partograph form is based on recording the developments observed during labor by specifying the time, and recording begins when the woman enters the active phase (cervical dilatation of 5-6 cm). This form not only shows the progress of the action, but also determines the deviation of the process from normal. In the partograph; There are three parameters that show the progress of birth, the health status of the baby and the health status of the mother. To determine the progress of labor; Cervical dilation, level of the baby's head, frequency and duration of uterine contractions in 10 minutes are monitored and recorded. To evaluate the baby's health status; The fetal heart rate (every 30 minutes), the presence of the amniotic membrane at each vaginal examination, the color of the fluid and the descent of the fetal head are evaluated and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Handan Guler, Assoc. Prof., Study Director — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)